CLINICAL TRIAL: NCT01317329
Title: "Reversibility of Cardiovascular Injury With Continuous Positive Airway Pressure (CPAP) Use: Mechanisms Involved"
Brief Title: "Reversibility of Cardiovascular Injury With CPAP Use: Mechanisms Involved"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K23HL094760 (NIH)
Record Dates: First submitted 2011-03-14; First posted 2011-03-17 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2015-09

CONDITIONS: Sleep Apnea, Obstructive; Hypoxia; Hypercapnia; Sleep Disorders; Obesity; Hypertension; Coronary Artery Vasospasm; Right Ventricular Overload; Left Ventricular Function Systolic Dysfunction; Ventricular Hypertrophy
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypoxia; Hypercapnia; Sleep Wake Disorders; Obesity; Hypertension; Coronary Vasospasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clinically prescribed CPAP therapy (Other): Clinically prescribed CPAP therapy
  Interventions: Other: Clinically prescribed CPAP therapy

INTERVENTIONS:
Other: Clinically prescribed CPAP therapy — CPAP as prescribed by attending physician

SUMMARY:
The purpose of this study is to determine the factors that are associated with improved cardiovascular function with the use of CPAP therapy on subjects diagnosed with moderate to severe obstructive sleep apnea.

DETAILED DESCRIPTION:
We will monitor non-invasively changes in arterial stiffness, cardiac mass, pulmonary pressures, endothelial function, etc. We will also assess the reversibility of these changes after only 5-7 days of not using the CPAP mask. In a subgroup of subjects we will explore changes in coronary flow response after 12 weeks of CPAP use compared with baseline.

ELIGIBILITY:
Inclusion Criteria:

* subjects naïve of CPAP therapy just recently diagnosed with moderate to severe obstructive sleep apnea (OSA). The degree of OSA is defined by results of a comprehensive polysomnogram requiring an apnea hypopnea index (AHI) >15 events/hour and Epworth score >10, or an AHI >20 events/hour
* either sex
* any race
* between 21-50 years old.

Exclusion Criteria:

* Systolic blood pressure >160 mmHg, or diastolic blood pressure >100 mmHg
* Changes in antihypertensive medications in the last 6 weeks
* Restless leg syndrome
* Average overnight oxygen saturation below 80%
* Current use of beta-blockers
* History of coronary artery disease
* History of Stroke
* Atrial fibrillation
* Peripheral vascular disease
* Suspected cardiac valve abnormality
* Ejection fraction <50%
* Type I and type II Diabetes Mellitus (DM)
* Asthma or confirmed Chronic Obstructive Pulmonary Disease
* Cigarette smoking in the last 6 months
* Raynaud's disease
* Pregnancy (the normal hormonal changes that occur in pregnancy affect greatly arterial stiffness parameters) If a subject becomes pregnant we will discontinue data collection.
* Physically incapable of resting on left lateral decubitus for 40 minutes.
* Mastectomy with lymph node removal that might preclude us to monitor blood pressures on both arms

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2011-03; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes in endothelium mediated response to brachial artery reactivity test between baseline and 4 and 12 weeks after CPAP therapy | 14 weeks
  Ultrasound based brachial artery reactivity tests will be performed at entry before CPAP therapy and at 4, 12 weeks post CPAP use and 5-7 days after CPAP withdrawal

SECONDARY OUTCOMES:
Changes in arterial stiffness between baseline and after CPAP treatment | 14 weeks
  Subjects will undergo pulse wave velocity testing with applanation tonometry. tonometry recordings will be at entry and after 4 and 12 weeks of CPAP use and 5-7- days after withdrawal.
Changes in coronary artery flow under a cold pressor test | 13 weeks
  A subset of subjects with abnormal endothelial function determined during the baseline scan and good echocardiographic images will be invited to participate on this portion of the test. We will record the response to a cold pressor test (submerging their hand in ice water for 1.5 minutes) on left anterior descending coronary artery velocities with transthoracic echocardiography at baseline and after 12 weeks of CPAP therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia E Korcarz, DVM, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Wisconsin Sleep, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Korcarz CE, Benca R, Barnet JH, Stein JH. Treatment of Obstructive Sleep Apnea in Young and Middle-Aged Adults: Effects of Positive Airway Pressure and Compliance on Arterial Stiffness, Endothelial Function, and Cardiac Hemodynamics. J Am Heart Assoc. 2016 Apr 3;5(4):e002930. doi: 10.1161/JAHA.115.002930. PMID 27039928